CLINICAL TRIAL: NCT01071772
Title: Metabolic Substrate Modulation in Insulin Treated Diabetics With and Without Heart Failure: The Effect of Hyperglycemia on Left Ventricular Function and Exercise Capacity.
Brief Title: The Effect of Hyperglycemia on LV Function and Exercise Capacity in Diabetics With and Without Heart Failure.
Acronym: METAMOD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Danish Heart Foundation (Other); Region midtjyllands sundhedsvidenskabelige forskningsfond (Unknown)
Responsible Party: Dr. Roni Ranghoej Nielsen, Dept. of cardiology, Aarhus University hospital, Skejby, Brendstrupgaardsvej 100, 8200 Aarhus N, Denmark
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: M20080151
Record Dates: First submitted 2010-02-16; First posted 2010-02-19 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-06

CONDITIONS: Heart Failure; Type 2 Diabetes
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus, Type 2 | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- euglycemia (Experimental)
  Interventions: Drug: insulin
- hyperglycemia (Experimental)
  Interventions: Drug: insulin

INTERVENTIONS:
Drug: insulin — There will be used individual intravenous insulin (actrapid) infusion to prevent non-intended hyperglycemia.

SUMMARY:
Diabetes and Heart Failure are diseases with high morbidity and increased risk of death. Former investigations has shown that diabetes worsens the prognosis of heart failure. However it is uncertain how short term diabetic dysregulation in type 2 diabetics affect cardiac function.

Our hypothesis is that short term dysregulation affects left ventricular function and exercise capacity in insulin treated type 2 diabetics with and without heart failure.

To elucidate this hypothesis diabetic patients with and without heart failure will be investigated after overnight state of either high or normal blood glucose levels on two separate occasions. Metabolic and hormonal parameters will be measured. Systolic and diastolic cardiac function will be assessed, exercise capacity and post exercise regional myocardial tissue velocity as well as 6 minutes walk test will be investigated on both occasions. The study will be a randomized cross-over design.

ELIGIBILITY:
Inclusion Criteria:

* Either normal ejection fraction (EF) or heart failure (EF =<45%)
* Insulin treated type 2

Exclusion Criteria:

* Forme stroke with significant physically or mentally disabilitating disorders
* advanced renal disease (creatinine levels >220 mM)
* advanced lever disease (alanine aminotransferase > 3 times over reference level).
* pregnancy
* other significant disabilitating disorders

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
1: Cardiac systolic (EF by 2D and 3D echocardiography) and diastolic (e´/E and E/A) function before and after exercise. | 1-4 weeks
Exercise capacity | 1-4 months

SECONDARY OUTCOMES:
Regional left ventricular function before and after maximum exercise(regional 2D tissue velocity and strain) | 1-4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hans Erik Boedker, Prof, MD, Study Director — Dept. of cardiolgy, Aarhus University hospital, Skejby. Brendstrupgaardsvej 100, 8200 Aarhus N, Denmark
Locations (1):
- Department ofCardiology, Aarhus University Hospital, Skejby, Aarhus, Central Jutland, Denmark